CLINICAL TRIAL: NCT00721448
Title: A Two-Cohort, Open-Label, Single and Multiple Dose Pharmacokinetic Study of 90 mg and 180 mg Doses of AZD6140 in Healthy Chinese Volunteers Living in China
Brief Title: An Open-Label, Single and Multiple Dose Pharmacokinetic Study of 90 mg and 180 mg Doses of AZD6140 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Marco Avila, AstraZeneca Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D5130C00054
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Pharmacokinetics
Keywords: Pharmacokinetics
MeSH Terms: interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AZD6140 — 90mg tablet, oral, once daily for the first day and twice daily from day 4 to 9
Drug: AZD6140 — 90 x 2 mg tablets, oral, once daily for the first day and twice daily from day 4 to 9

SUMMARY:
This will be a single centre study conducted at the 3rd hospital affiliated to Peking University. Approximately 24 healthy Chinese volunteers, male and female, will be recruited to obtain at least 20 evaluable volunteers. The primary objective of this study is to characterize the pharmacokinetics of AZD6140 and its active metabolite AR-C124910XX after single and multiple (twice daily) doses of AZD6140 90 mg and 180 mg in healthy Chinese volunteers. The secondary objective of this study is to determine the safety and tolerability of single and multiple (twice daily) 90 mg and 180 mg doses of AZD6140 by physical examination, clinical laboratory tests, vital signs, and collection of adverse events in healthy Chinese volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Chinese ethnicity defined as having both parents and 4 grandparents who are Chinese
* Have a normal Body size and weigh at least 50 kg

Exclusion Criteria:

* History of diseases or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs determined by the investigator
* Current and/or past history of intolerance or hypersensitivity to drugs with a similar chemical structure or mechanism of action to AZD6140 or any ingredient in its formulation
* Symptoms of any clinically significant illness within 2 weeks of screening
* A personal or family history of bleeding diatheses or a reasonable suspicion of vascular abnormalities including aneurysms

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
AZD6140 and AR-C124910XX concentration | -2,0,0.5,1,2,3,4,6,8,12,18,24,36,48,72 hours on days 4,5,6,7,8and 9. Day 10 the samples are at the specified timeframes (0,0.5,1,2,3,4,6,8,12,18,24,36,48,72 hours)

SECONDARY OUTCOMES:
determine the safety and tolerability of single and multiple doses of AZD6140 by physical examination, clinical laboratory tests, vital signs, and collection of adverse events | day -1, 4, 7, 10, 13+3~5

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Gillette, Study Director — AZ Pharmaceuticals - US; Li Haiyan, MD, Principal Investigator — 3rd hospital affiliated to Peking University
Locations (1):
- Research Site, Beijing, China

REFERENCES:
- [Derived] Li H, Butler K, Yang L, Yang Z, Teng R. Pharmacokinetics and tolerability of single and multiple doses of ticagrelor in healthy Chinese subjects: an open-label, sequential, two-cohort, single-centre study. Clin Drug Investig. 2012 Feb 1;32(2):87-97. doi: 10.2165/11595930-000000000-00000. PMID 22168538